CLINICAL TRIAL: NCT06955676
Title: The Effects of Moderate Intensity, Time-matched Cycle Ergometer vs. Treadmill Exercise Training on Parameters Associated With Physiological Resilience in Older Adults: A Pilot Study
Brief Title: The Effects of Moderate Intensity Cycle Ergometer vs. Treadmill Training on Physiological Resilience in Older Adults
Acronym: MICeT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Principal Investigator, Bethan Phillips, Professor of Translational Physiology, University of Nottingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMHS 367-0923
Record Dates: First submitted 2024-09-27; First posted 2025-05-02 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2024-09

CONDITIONS: Older People
Keywords: aerobic exercise; older adults; elderly; resilience; treadmill; cycle ergometer

STUDY DESIGN:
Intervention Model Description: Group 1: moderate-intensity treadmill training Group 2: moderate-intensity cycle ergometer training Group 3: control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- treadmill exercise (Experimental): All participants should visit the research unit and attend the sessions 3 times a week for 5 weeks. Participants in this group will conduct moderate-intensity (64-76% of Heart rate maximum) treadmill training for 40 minutes each session. There is a 5-min warm-up before the intervention and a 5-min cool-down period after the intervention.
  Interventions: Other: treadmill exercise
- cycle ergometer exercise (Experimental): All participants should visit the research unit and attend the sessions 3 times a week for 5 weeks. Participants in this group will conduct moderate-intensity (64-76% of Heart rate maximum) cycle ergometer training for 40 minutes each session. There is a 5-min warm-up before the intervention and a 5-min cool-down period after the intervention.
  Interventions: Other: cycle ergometer exercise
- control group (No Intervention): The control group will receive 'no intervention'.

INTERVENTIONS:
Other: treadmill exercise — Intervention consists of exercises only. Participants in this group will walk on a treadmill. The heart rates of the participants will be monitored with a heart rate monitor while exercising in order to maintain moderate-intensity.
  Arms: treadmill exercise
Other: cycle ergometer exercise — Intervention consists of exercises only. Participants in this group will cycle on an ergometer. The heart rates of the participants will be monitored with a heart rate monitor while exercising in order to maintain moderate-intensity.
  Arms: cycle ergometer exercise

SUMMARY:
Government guidelines suggest that we should all take part in approximately two and a half hours each week of moderate-intensity aerobic exercise. Older adults are particularly important as their overall health may decline as they get older. Therefore, exercising is important especially for older adults to improve heart and muscle health and functioning in carrying out tasks of daily living. The overall effects of aging on the body can make people less likely to withstand challenges to the body - this is termed 'resilience'. Although aerobic exercise is not super easy and requires continuity, it is not extremely difficult to get used to. However, we still do not know if some types of aerobic exercise are better for you than others at improving resilience. Therefore, this study will look at cycling vs walking to see if one is better at improving resilience in older adults who are 60-80 years old. You will be trained on either a treadmill or cycle ergometer and these exercise sessions will be done over 5 weeks, 3 days a week. Each session will last 40 minutes, start with warm-up and end with cool-down sessions. Assessments will include heart, lung, muscle, and memory and thinking measurements, all of which will be taken before and after the intervention period. This work will help us to better understand how we can improve exercise prescriptions for older adults to sustain their health and functioning in their daily life.

DETAILED DESCRIPTION:
Physiological resilience refers to the capacity to retain or regain physical function in the presence of diseases or age-related impairments. Poor resilience may increase vulnerability to stress, which could lead to negative functional and clinical consequences like a prolonged course of illness/hospitalization, reduced physical activity, an elevated risk of frailty, and even mortality. Physiological resilience is particularly crucial because it declines, and the likelihood of many stresses rises with age. Therefore, it is important to promote older populations' physiological resilience reserves and resources (increase their readiness levels against potential future stressors that are more likely to be seen when an individual gets older). Since risk of having stressors increases with advanced age, there is a relationship between aging and reduced readiness to stressors (low physiological resilience).

The scientific data establishing the beneficial effects of exercise is undeniable, and the advantages of exercise considerably outweigh the hazards in most adults. Although the existing evidence supports that exercise interventions are a potent tool to foster resilience in older adults, there is still a need of future studies regarding this information. Aerobic exercise (AE), one of the most recommended exercise types by the literature, has also been stated as a beneficial tool to promote physiological resilience at all stages of life through increased growth factor expression and neuroplasticity, which lower the destructive effects of chronic stress. Also, aerobic fitness has been shown to be one of the best predictors of resilience. Government guidelines recommend performing moderate-intensity AE 150 minutes per week. However, the literature does not elaborate on the details of AE interventions on physiological resilience and there is a lack of information on which AE modality is better for this purpose. Although the literature supports the idea of AE being a beneficial tool to improve health and physical fitness goals as well as resilience, it can clearly be seen that there is a need for future research regarding both the comparison of AE modalities in older adults and the effects of AE intervention to promote physiological resilience. Thus, this study will be the first to compare the effects of moderate intensity time-matched AE modalities (cycle ergometer versus treadmill training versus control group) on the parameters associated with physiological resilience (muscle mass/strength, cognition, dexterity, functional ability, cardiorespiratory fitness, and neuromuscular function) in older adults. The intervention period will last 5 weeks, 3 days a week, with 40-minute sessions. The research question will be 'Which AE modality is better in improving determinants of physiological resilience?'. This work will allow us to understand the relationship between AE and physiological resilience in a more detailed way and to prescribe better exercise prescriptions in the future.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study
* Participants who are able to perform exercises safely and freely
* Participants who are 60-80 years old

Exclusion Criteria:

* Cardiopulmonary diseases except for well-controlled hypertension and asthma
* Severe cognitive impairment
* Joint disorders avoiding exercise participation
* A recent heart attack, unstable angina, or severe heart failure
* Having taken part in a research study in the last 3 months involving invasive procedures or an inconvenience allowance
* Participants who are currently engaging in more than 150 min of moderate-intensity exercise per week or 75 min of vigorous-intensity exercise per week (WHO physical activity recommendations)

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
The change in vastus lateralis mass | at baseline (pre-intervention) and at the week 5 (post-intervention)
  Bioelectrical impedance analysis (BIA) and ultrasound will be used for this. Muscle thickness, fascicle length, and pennation angle will be measured on ultrasound. BIA is simple to use, places a minimal burden on individuals, uses lightweight and inexpensive equipment, and, most significantly, provides no radiation risk compared to many other methods. It is also found feasible and reliable for the measurement of muscle mass for adults in clinical settings. Ultrasonography is also a technology that is portable, safe, and clearly distinguishes between muscle and subcutaneous fat tissues as well as a valid and novel tool for muscle mass assessment.
The changes of muscle strength with maximum voluntary contraction of knee extension | at baseline (pre-intervention) and at the week 5 (post-intervention)
  Maximum voluntary contraction is a standardized technique for assessing muscle strength in healthy older adults. Knee extension strength will be measured with an isometric dynamometer.
The change in cardiorespiratory fitness (CRF) capacity via the Ekblom-bak (EB) test | at baseline (pre-intervention) and at the week 5 (post-intervention)
  The EB-test consists of exercise at one standardized, low work rate followed by a higher, individually set work rate. Both work rates are performed for 4 minutes at a cadence of 60rpm on a cycle ergometer. The individual higher work rate is chosen by the researcher according to the participants' gender, age, and training background. The higher work rate aims to reach the Borg rate of perceived exertion (RPE) 12-16. Heart rate is measured during the last minute of each work rate (at 3:15, 3:30, 3:45, and 4:00). Then, VO2max is estimated with a formula.
The difference in neuromuscular function via force accuracy task | at baseline (pre-intervention) and at the week 5 (post-intervention)
  Force accuracy is an important parameter since most daily activities are conducted at submaximal levels, where force fluctuation can be observed and reduce the ability to create an intended movement. Force accuracy will be measured on OTBiolab+ application.
The changes in functional ability via the Timed Up and Go test (TUG) | at baseline (pre-intervention) and at the week 5 (post-intervention)
  The TUG is a tool for assessing lower limb functional ability and its use has been recommended by the literature. The time required to finish the test is commonly utilised as the primary outcome of the evaluation. This test has previously been used in several studies to assess functional ability.
The difference between upper limb dexterity time before and after the intervention via 9-hole peg task | at baseline (pre-intervention) and at the week 5 (post-intervention)
  The 9-hole peg test has been shown to be a valid and reliable tool to measure upper extremity dexterity in various groups including healthy older adults. The number of seconds it takes for the participant to complete the test is used for scoring. A shorter completion time is a better value.
The changes in cognitive function via Mini-ACE | at baseline (pre-intervention) and at the week 5 (post-intervention)
  The Mini-ACE is a brief cognitive screening test that evaluates four main cognitive areas (orientation, memory, language and visuospatial function). Higher value on this scale means better cognition.
The changes of muscle strength with handgrip strength | at Baseline (pre-assessment) and at the week 5 (post-assessment)
  Isometric hand grip strength is closely correlated with the strength of the muscles in the lower extremities, and the torque of the knee, and poor mobility is clinically indicated by low handgrip strength. Higher values mean better results.
The change in cardiorespiratory fitness (CRF) capacity via 6-minute walking test (6MWT) | at baseline (pre-intervention) and at the week 5 (post-intervention)
  In the 6MWT, participants walk as much as they can for six minutes along a continuous, interior track that is 30 metres long and has a hard surface. It is a simple, cost-effective, and validated tool in several populations, and it has been frequently used to measure CRF as a field test. The distance covered on this test is reported. A higher distance covered means a better result.
The difference in neuromuscular function via balance time in The Short Physical Performance Battery (SPPB) on motion platform | at baseline (pre-intervention) and at the week 5 (post-intervention)
  Balance will be measured on FootScan (centre of pressure, distance travelled, ellipse area).
The changes in functional ability via Short Physical Performance Battery Test | at baseline (pre-intervention) and at the week 5 (post-intervention)
  Short Physical Performance Battery test includes the chair rise, balance, walk and gait speed assessments for functional mobility. An overall score is determined on a scale from 0 to 12, with lower scores representing a more severe level of disability and higher scores representing more functionally normal levels.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet C Yildirim, PhD, Study Director — The University of Nottingham
Locations (1):
- The University of Nottingham/Medical School, Derby, Derbyshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Whitson HE, Duan-Porter W, Schmader KE, Morey MC, Cohen HJ, Colon-Emeric CS. Physical Resilience in Older Adults: Systematic Review and Development of an Emerging Construct. J Gerontol A Biol Sci Med Sci. 2016 Apr;71(4):489-95. doi: 10.1093/gerona/glv202. Epub 2015 Dec 29. PMID 26718984
- [Background] Hadley EC, Kuchel GA, Newman AB; Workshop Speakers and Participants. Report: NIA Workshop on Measures of Physiologic Resiliencies in Human Aging. J Gerontol A Biol Sci Med Sci. 2017 Jul 1;72(7):980-990. doi: 10.1093/gerona/glx015. PMID 28475732
- [Background] Cosco TD, Howse K, Brayne C. Healthy ageing, resilience and wellbeing. Epidemiol Psychiatr Sci. 2017 Dec;26(6):579-583. doi: 10.1017/S2045796017000324. Epub 2017 Jul 6. PMID 28679453
- [Background] Sampedro-Piquero P, Moreno-Fernandez RD. Building Resilience with Aerobic Exercise: Role of FKBP5. Curr Neuropharmacol. 2021;19(8):1156-1160. doi: 10.2174/1570159X19666210408124937. PMID 33829973
- [Background] Arida RM, Teixeira-Machado L. The Contribution of Physical Exercise to Brain Resilience. Front Behav Neurosci. 2021 Jan 20;14:626769. doi: 10.3389/fnbeh.2020.626769. eCollection 2020. PMID 33584215
- [Background] Lee SY, Ahn S, Kim YJ, Ji MJ, Kim KM, Choi SH, Jang HC, Lim S. Comparison between Dual-Energy X-ray Absorptiometry and Bioelectrical Impedance Analyses for Accuracy in Measuring Whole Body Muscle Mass and Appendicular Skeletal Muscle Mass. Nutrients. 2018 Jun 7;10(6):738. doi: 10.3390/nu10060738. PMID 29880741
- [Background] Mijnarends DM, Meijers JM, Halfens RJ, ter Borg S, Luiking YC, Verlaan S, Schoberer D, Cruz Jentoft AJ, van Loon LJ, Schols JM. Validity and reliability of tools to measure muscle mass, strength, and physical performance in community-dwelling older people: a systematic review. J Am Med Dir Assoc. 2013 Mar;14(3):170-8. doi: 10.1016/j.jamda.2012.10.009. Epub 2012 Dec 29. PMID 23276432
- [Background] Scott JM, Martin DS, Ploutz-Snyder R, Matz T, Caine T, Downs M, Hackney K, Buxton R, Ryder JW, Ploutz-Snyder L. Panoramic ultrasound: a novel and valid tool for monitoring change in muscle mass. J Cachexia Sarcopenia Muscle. 2017 Jun;8(3):475-481. doi: 10.1002/jcsm.12172. Epub 2017 Jan 3. PMID 28052593
- [Background] Meldrum D, Cahalane E, Conroy R, Fitzgerald D, Hardiman O. Maximum voluntary isometric contraction: reference values and clinical application. Amyotroph Lateral Scler. 2007 Feb;8(1):47-55. doi: 10.1080/17482960601012491. PMID 17364436
- [Background] Lauretani F, Russo CR, Bandinelli S, Bartali B, Cavazzini C, Di Iorio A, Corsi AM, Rantanen T, Guralnik JM, Ferrucci L. Age-associated changes in skeletal muscles and their effect on mobility: an operational diagnosis of sarcopenia. J Appl Physiol (1985). 2003 Nov;95(5):1851-60. doi: 10.1152/japplphysiol.00246.2003. PMID 14555665
- [Background] Dourado VZ, Nishiaka RK, Simoes MSMP, Lauria VT, Tanni SE, Godoy I, Gagliardi ART, Romiti M, Arantes RL. Classification of cardiorespiratory fitness using the six-minute walk test in adults: Comparison with cardiopulmonary exercise testing. Pulmonology. 2021 Nov-Dec;27(6):500-508. doi: 10.1016/j.pulmoe.2021.03.006. Epub 2021 May 4. PMID 33958319
- [Background] Santana MG, de Lira CA, Passos GS, Santos CA, Silva AH, Yoshida CH, Tufik S, de Mello MT. Is the six-minute walk test appropriate for detecting changes in cardiorespiratory fitness in healthy elderly men? J Sci Med Sport. 2012 May;15(3):259-65. doi: 10.1016/j.jsams.2011.11.249. Epub 2011 Dec 11. PMID 22154397
- [Background] Singh NB, Arampatzis A, Duda G, Heller MO, Taylor WR. Effect of fatigue on force fluctuations in knee extensors in young adults. Philos Trans A Math Phys Eng Sci. 2010 Jun 13;368(1920):2783-98. doi: 10.1098/rsta.2010.0091. PMID 20439273
- [Background] Cruz-Jentoft AJ, Baeyens JP, Bauer JM, Boirie Y, Cederholm T, Landi F, Martin FC, Michel JP, Rolland Y, Schneider SM, Topinkova E, Vandewoude M, Zamboni M; European Working Group on Sarcopenia in Older People. Sarcopenia: European consensus on definition and diagnosis: Report of the European Working Group on Sarcopenia in Older People. Age Ageing. 2010 Jul;39(4):412-23. doi: 10.1093/ageing/afq034. Epub 2010 Apr 13. PMID 20392703
- [Background] Gojanovic M, Holloway-Kew KL, Hyde NK, Mohebbi M, Shivappa N, Hebert JR, O'Neil A, Pasco JA. The Dietary Inflammatory Index Is Associated with Low Muscle Mass and Low Muscle Function in Older Australians. Nutrients. 2021 Apr 1;13(4):1166. doi: 10.3390/nu13041166. PMID 33916033
- [Background] Przkora R, Kinsky MP, Fisher SR, Babl C, Heyde CE, Vasilopoulos T, Kaye AD, Volpi E. Functional Improvements Utilizing the Short Physical Performance Battery (SPPB) in the Elderly after Epidural Steroid Injections. Curr Pain Headache Rep. 2019 Feb 22;23(2):14. doi: 10.1007/s11916-019-0748-2. PMID 30796532